CLINICAL TRIAL: NCT04649164
Title: Learning to PERSEVERE: Peer Mentor Support and Caregiver Education in Lewy Body Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20030604; 5P30AG064200-02 (NIH)
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Lewy Body Disease; Parkinson Disease Dementia; Dementia With Lewy Bodies
Keywords: caregiver strain; caregiving mastery; peer mentor; caregiver education; Lewy Body Disease; Parkinson's Disease; social support
MeSH Terms: conditions — Lewy Body Disease; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Focus group participants (Other): Subjects participating in focus groups will be either:
  1. caregiver mentees in our previous peer mentoring study
  2. peer mentors and completed 16 weeks of mentoring in our previous peer mentoring study
  3. current family caregivers of community-dwelling LBD patients in the Chicago area.
  The investigators will conduct virtual focus groups using a password-protected videoconference platform. The informed consent process will take place online prior to the focus group. Focus groups will be led by a qualified neuropsychologist using open-ended questions. The aim of these groups is to revise and improve upon our previous peer mentor program's curriculum. Participants will be presented with the previous program's curriculum and a variety of proposed educational resources for inclusion in the revised curriculum. The investigators will obtain participants' feedback. Focus groups will be recorded and transcribed.
  Interventions: Other: Focus group to provide feedback on educational materials and mentoring program
- Peer mentors (Other): Mentors will attend one 6-7 hour virtual training session. Study expectations and logistics will be reviewed with each potential mentor prior to the training session via phone. Informed consent process will take place online via REDCap prior to the training session. Baseline data will be collected via online surveys. Next, mentors will receive training regarding topics including active listening, mentoring, goal-and boundary-setting, an overview of LBD, risk factors for hospitalization, impact on caregiver, practical approaches to symptom management, and caregiving issues. The study team will present the PERSEVERE curriculum and accompanying handbook. The team will solicit questions and lead roleplay conversations. Finally mentors will complete post-training assessments. Once all caregiver mentees (Arm 3) are recruited, the mentors will contact their mentees once weekly by phone for 16 weeks to deliver the PERSEVERE curriculum.
  Interventions: Behavioral: Peer mentor support and caregiver intervention
- Caregiver mentees (Experimental): Once Aim 2 is complete and mentors have been trained, caregiver mentees will be matched with mentors by relationship to LBD patient, then by sex and age, as much as possible. The study team will contact mentees once a match is available for them. The mentee will complete baseline primary and secondary outcome assessments online via REDCap, including: mastery and loneliness scales, Short Zarit Burden Interview, Hospital Anxiety and Depression Scale. The team will provide the mentor's contact information and send the PERSEVERE handbook. Mentoring pairs will begin the 16-week peer mentor program. Pairs will be expected to speak for >15-30 minutes weekly, and to review that week's PERSEVERE topics in the handbook before or during each call to facilitate meaningful conversations. Mentors and mentees will complete online study diaries every 2 weeks. Upon completion of the 16-week mentor program, mentors and mentees will be sent a link to complete postmentoring assessments online.
  Interventions: Behavioral: Peer mentor support and caregiver intervention

INTERVENTIONS:
Behavioral: Peer mentor support and caregiver intervention — Sixteen-week modular curriculum with printed/online workbook, additional resources, and weekly phone discussion with Lewy Body Dementia peer mentor.
  Arms: Caregiver mentees; Peer mentors
Other: Focus group to provide feedback on educational materials and mentoring program — Participation in a 2-3 hour focus group to review pilot and revised materials and provide feedback
  Arms: Focus group participants

SUMMARY:
The investigators propose to adapt, improve, and implement a peer mentor support and caregiver education (PERSEVERE) program to improve LBD-specific caregiving mastery. Lewy body dementia (LBD) is the second most common dementia, comprising Parkinson's Disease (PD) dementia and Dementia with Lewy Bodies. LBD causes deterioration in multiple cognitive, motor, and neuropsychiatric domains, leading to heavy reliance on family caregivers. Patients with LBD are at a far greater risk of hospitalizations for falls, neuro-psychiatric symptoms, and infections, which are often preventable or treatable at home if recognized. Studies cite a crucial need for education and support of LBD caregivers, who face high rates of caregiver strain and adverse outcomes. Evidence from other chronic conditions supports peer mentoring as a potentially effective intervention to provide education and social support. PERSEVERE builds on our team's ongoing work of creating and testing a peer mentoring program for homebound PD patients' caregivers that has shown promising feasibility and acceptability. In the proposed project, the investigators will convene focus groups of former mentors and mentees, along with current caregivers, to provide formative information to shape the revised PERSEVERE curriculum that will include in-person mentor training and a comprehensive mentoring handbook. The curriculum will focus on key areas of LBD caregiving mastery, including: fall prevention, infections, neuropsychiatric symptoms (particularly hallucinations, delusions, anxiety, and depression), and advance directives. The investigators will enroll and train a new cohort of 36 LBD caregiver peer mentors who will be matched with 30 current LBD caregivers. Each pair will be instructed to speak on a weekly basis, using the 16-week structured curriculum as a framework. The study team will support the mentors with monthly conference calls and day-to-day availability for concerns. The investigators will assess the feasibility and fidelity of the intervention via online study diaries tracking the frequency, duration, and content of calls. During mentor training, the investigators will assess the change in mentors' caregiver mastery and LBD knowledge pre- and post-training. During the PERSEVERE intervention, the investigators will determine the change in mentees' caregiver mastery, LBD knowledge, and loneliness.

DETAILED DESCRIPTION:
Scientific Premise. PERSEVERE is a theory-based intervention that applies Social Cognitive Theory constructs to the revised Stress Process Model to improve caregiving mastery and ultimately, outcomes. PERSEVERE targets education about common causes of hospitalization in LBD patients combined with social support from trained peer mentors to enhance caregivers' mastery and LBD knowledge. Social Cognitive Theory (SCT) proposes that behavior change is dynamic, affected by expectations, observational learning, and reciprocal influences from the environment.

Study procedures. Aim 1 (Fall 2020): Revise the mentor training curriculum, conversation guides, and resource handbook. The team will convene focus groups of previously trained mentors, LBD caregivers, and LBD professionals, present each group with the original mentor curriculum (training presentation slides and handbook) and the proposed educational resources for inclusion in the revised curriculum and obtain their feedback. Framework analysis will be used to guide the revision of the mentoring curriculum, with provision of practical checklists, goal setting, and step-by-step guides for key areas of LBD caregiving mastery in addition to social support, structured as the 16-week PERSEVERE curriculum.

Aim 2 (Winter 2021): Recruit and screen 36 peer mentors as PERSEVERE is being revised, followed by two 6-7 hour training sessions for mentors in early 2021. Each selected mentor will attend one training session, where the following content will be delivered: 1) study logistics, expectations, and informed consent; 2) baseline mentor data collection; 3) active listening, mentoring, goal- and boundary-setting; 4) overview of LBD, risk factors for hospitalization, impact on caregiver; and 5) practical approaches to symptom management and caregiving issues. The week-by-week PERSEVERE curriculum will be presented along with the accompanying handbook. The investigators will solicit questions and role-play conversations. The study team will encourage mentors to direct their mentees to call their respective medical teams with specific medical questions, however the study team will inform the mentors that they may contact the study team directly for non-emergent advice and resources. Mentors will complete post-training assessments and will receive a training stipend. Mentors' caregiver mastery will be assessed using Pearlin and Schooler's scale pre- and post-training.

Aim 3 (Spring-Summer 2021): Recruit 30 LBD caregivers and conduct baseline assessments including demographics, relationship to LBD patient, and duration of caregiving. Mentors will be matched to caregivers by relationship to LBD patient, then by sex and age, as much as possible. Mentor-mentee pairs will be formed and the PERSEVERE handbook and contact information will be distributed. Pairs will be expected to speak for >15-30 minutes weekly, and to review that week's PERSEVERE topics in the handbook before or during each call to facilitate meaningful conversations. Discussions are not scripted and will not necessarily be limited to that week's topics. Mentors and mentees will complete online study diaries every 2 weeks, assessing intervention fidelity. Up to 3 reminders will be sent to complete each study diary, and if missing, a team member will call the participant(s). Mentors will participate in a total of 4 recorded monthly conferences with the study team. Mentees' caregiver mastery, strain, anxiety, and depression will be assessed at baseline and after the 16-week program. Feasibility will be assessed via online surveys and study team phone call follow-up.

This pilot study will determine the necessary qualities of mentors and matching, the content of the mentor training and PERSEVERE handbook, and the effect sizes of the intervention to determine the sample size for a forthcoming R01.

ELIGIBILITY:
Inclusion Criteria:

1. Focus group participants

   1. Each subject must be 21 years of age or older. A subject may identify as any sex, any race, and any ethnicity.
   2. Subjects must be either:

   i. Individuals who served as peer mentors in our previous study of caregiver peer mentoring and completed at least 16 weeks of mentoring. ii. Individuals who were caregiver mentees in our previous study of caregiver peer mentoring who completed 16 weeks of mentoring. iii. Current informal family caregivers of community-dwelling LBD patients in the Chicago area, recruited from Rush University System for Health and Advocate Aurora Health, who have not participated in mentoring. c. Each subject must be primarily English-speaking. d. Each subject must be willing and able to attend a virtual, online focus group via an internet- and video-camera-equipped computer, tablet, or smartphone.
2. Peer mentors

   1. Each subject must be 21 years of age or older. A subject may identify as any sex, any race, and any ethnicity.
   2. Each subject must be a non-professional caregiver (defined as cohabitating with or spending >10 hours weekly on unpaid caregiving duties) of LBD patients. Mentors may participate regardless of their loved one's status (living at home, institutionalized, or deceased).

   i. If mentors also receive compensation for a portion of their time spent on caregiving duties through state or community programs, they may participate as long as they cohabitate or spend >10 hours providing unpaid care to their loved one. c. Each subject must have >2 years of LBD caregiving experience d. Each subject must be primarily English-speaking. e. Each subject must have a working email address and internet access. f. Each subject must have a working telephone number at which he or she can be reached and which he or she is willing to share with the matched mentee.

   g. Each subject who will attend an online peer mentor training session must have an internet- and video-camera-equipped computer, tablet, or smartphone
3. Caregiver mentees

   1. Each subject must be 21 years of age or older. A subject may identify as any sex, any race, and any ethnicity.
   2. Each subject must be a non-professional, unpaid caregiver, as defined above, of a community-dwelling LBD patient.
   3. Each subject must be interested in improving their caregiving mastery.
   4. Each subject must be primarily English-speaking.
   5. Each subject must have a working email address and internet access.
   6. Each subject must have a working telephone number at which he or she can be reached and which he or she is willing to share with the matched mentor.

Exclusion Criteria:

1. Subjects exhibiting symptoms of a severe psychiatric disorder interfering with their ability to participate in the study, as determined by a study team member or the PI.
2. Subjects who are primarily non-English-speaking.
3. Terminal illness (life expectancy of < 12 months).

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jori E Fleisher, MD MSCE, Principal Investigator — Rush University Medical Center, Department of Neurological Scienecs
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fleisher JE, Suresh M, Levin ME, Hess SP, Akram F, Dodson D, Tosin M, Stebbins GT, Woo K, Ouyang B, Chodosh J. Learning to PERSEVERE: A pilot study of peer mentor support and caregiver education in Lewy body dementia. Parkinsonism Relat Disord. 2023 Aug;113:105492. doi: 10.1016/j.parkreldis.2023.105492. Epub 2023 Jun 24. PMID 37385161

RESULTS

PARTICIPANT FLOW:
Groups:
- Focus Group Participants: Subjects participating in focus groups will be either:
  1. caregiver mentees in our previous peer mentoring study
  2. peer mentors and completed 16 weeks of mentoring in our previous peer mentoring study
  3. current family caregivers of community-dwelling LBD patients in the Chicago area.
  The investigators will conduct virtual focus groups using a password-protected videoconference platform. The informed consent process will take place online prior to the focus group. Focus groups will be led by a qualified neuropsychologist using open-ended questions. The aim of these groups is to revise and improve upon our previous peer mentor program's curriculum. Participants will be presented with the previous program's curriculum and a variety of proposed educational resources for inclusion in the revised curriculum. The investigators will obtain participants' feedback. Focus groups will be recorded and transcribed.
  Focus group to provide feedback on educational materials and mentoring program: Participation in a 2-3 hour focus group to review pilot and revised materials and provide feedback
Period: Overall Study
Arm/Group | Focus Group Participants | Peer Mentors | Caregiver Mentees
Started | 19 | 36 | 32
Completed | 18 | 35 | 28
Not Completed | 1 | 1 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Participant's care recipient expired | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Focus Group Participants | Peer Mentors | Caregiver Mentees | Total
Number analyzed (Participants) | 19 | 36 | 32 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 15 | 12 | 30
  >=65 years | 16 | 21 | 20 | 57
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [67 to 77] | 66 [62 to 73] | 68 [61.5 to 71] | 68 [62 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 34 | 30 | 82
  Male | 1 | 2 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 18 | 35 | 29 | 82
  Unknown or Not Reported | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 17 | 33 | 29 | 79
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 19 | 36 | 32 | 87

OUTCOME MEASURES:

1. Primary Outcome: Mastery Scale
Description: A 7-item scale measuring the extent to which a participant sees life as being under his/her personal control vs. something that is fatalistically ruled. Scores range from 7 to 28, with higher scores indicating greater levels of mastery
Time Frame: Pre- and post-mentor training; pre- and post-mentoring intervention for mentees (16 weeks)
Population: 35 mentors trained; we intentionally overrecruited peer mentors in order to ensure an adequate number of mentors who could be matched with caregiver mentees. We matched each of 30 mentees with one mentor, such that 5 mentors were trained but did not complete the 16 weeks of mentoring (effectively, "backup" mentors). This outcome was NOT assessed in the focus group arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentors | Caregiver Mentees
Number analyzed (Participants) | 30 | 28
units on a scale
  Pearlin Mastery Score (mean) at baseline | 21.65 (3.09) | 18.91 (2.90)
  Pearlin Mastery Score (mean) at week 16 of mentoring | 22.13 (3.47) | 19.2 (2.95)
Statistical Analysis 1: Comparison: Peer Mentors vs Caregiver Mentees; Paired t-tests comparing peer mentors' baseline and 16-week scores, and caregiver mentees' baseline and 16-week scores, respectively; Test type: Superiority; p = 0.36, t-test, 2 sided

2. Secondary Outcome: Loneliness Scale
Description: A 3-item, validated measurement of a participant's feelings of isolation or disconnectedness. Scores can range from 3-9, with higher scores indicating greater loneliness
Time Frame: pre- and post-mentoring intervention for mentees (16 weeks)
Population: As pre-specified, this measure was only gathered in caregiver mentees. Neither focus group participants nor mentors answered this scale. Two of 30 mentees did not complete the 16-week visit, and therefore 28/30 mentees had data available at both baseline AND 16 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver Mentees
Number analyzed (Participants) | 28
units on a scale
  Baseline | 5.64 (1.99)
  16 weeks (post-intervention) | 5.71 (2.16)

3. Secondary Outcome: Short Zarit Burden Interview (ZBI-12)
Description: A 12-item, validated measurement of caregiver burden in older adults. Scores range from 0-48, with higher scores indicating greater caregiver burden
Time Frame: pre- and post-mentoring intervention for mentees (16 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Mentees
Number analyzed (Participants) | 28
score on a scale
  Baseline | 23.18 (8.25)
  Week 16 (post-intervention) | 22.18 (8.52)
Statistical Analysis 1: Comparison: Caregiver Mentees; Test type: Superiority; p = 0.30, t-test, 2 sided

4. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) - Anxiety Score
Description: Anxiety subscale of the Hospital Anxiety and Depression Scale, where seven items measure anxiety. Total possible subscale range 0-21, where higher scores indicate worse outcome/more anxiety. A score >8 on the subscale indicates probable symptoms
Time Frame: 16 weeks
Population: As pre-specified, we analyzed only caregiver mentee participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Mentees
Number analyzed (Participants) | 28
score on a scale
  Baseline | 9.5 (4.18)
  16 weeks | 8.79 (3.78)
Statistical Analysis 1: Comparison: Caregiver Mentees; Test type: Superiority; p = 0.1, t-test, 2 sided

5. Secondary Outcome: Geriatric Depression Scale - Short Form (GDS-SF)
Description: Brief, 15-item, highly validated scale for measuring depression in older adults, total possible range of 0-15, where a score >5 suggests depression
Time Frame: 16 weeks
Population: As pre-specified, we gathered and analyzed this outcome in caregiver mentees only. 28/30 mentees completed both baseline and 16-week assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Mentees
Number analyzed (Participants) | 28
score on a scale
  Baseline | 5.0 (3.76)
  16 weeks | 4.22 (3.19)
Statistical Analysis 1: Comparison: Caregiver Mentees; Test type: Superiority; p = 0.04, t-test, 2 sided; Mean Difference (Final Values) = .78

6. Secondary Outcome: Dementia Attitudes Scale (DAS)
Description: A validated, 20-item scale measuring participants' attitudes toward dementia and individuals with dementia. Scores can range from 7-140, with higher scores indicating more positive attitudes
Time Frame: pre- and post-mentoring intervention for mentees (16 weeks)
Population: This outcome was not assessed in the focus group arm, as pre-specified.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Mentors | Caregiver Mentees
Number analyzed (Participants) | 30 | 28
score on a scale
  Baseline | 120.97 (11.76) | 104.25 (13.58)
  16 weeks (post-intervention) | 121.60 (11.81) | 111.57 (9.38)

7. Secondary Outcome: Duration of Mentoring Calls
Description: Online structured survey of mentoring phone call duration, in minutes
Time Frame: Assessed at weeks 2, 4, 6, 8, 10, 12, 14, 16; average value calculated at week 16
Population: As pre-specified, only mentees' reported call duration was analyzed. 28/30 mentees completed the intervention and week 16 surveys.
Measure: Median (Full Range); unit: minutes
Arm/Group | Caregiver Mentees
Number analyzed (Participants) | 28
minutes | 45.04 [12 to 138.75]

8. Secondary Outcome: Hospital Anxiety and Depression Scale - Depression Score
Description: Depression subscale of the Hospital Anxiety and Depression Scale, where seven items measure depression. Total possible subscale range 0-21, where higher scores indicate worse outcome/more depression. A score >8 on the subscale indicates probable symptoms
Time Frame: 16 weeks
Population: As pre-specified, only caregiver mentees completed this measure at baseline and 16 weeks, with 28 total mentees completing the measure at both time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Mentees
Number analyzed (Participants) | 28
score on a scale
  Baseline | 6.32 (3.4)
  16 weeks | 5.61 (3.5)
Statistical Analysis 1: Comparison: Caregiver Mentees; Test type: Superiority; p = 0.13, t-test, 2 sided

9. Other Pre Specified Outcome: Frequency of Mentoring Calls
Description: Online structured survey of number of calls
Time Frame: Assessed at 2, 4, 6, 8, 10, 12, 14, and 16 weeks; summed total phone calls at week 16 reported
Population: As pre-specified, only caregiver mentees' responses were analyzed for call frequency.
Measure: Median (Full Range); unit: phone calls
Arm/Group | Caregiver Mentees
Number analyzed (Participants) | 28
phone calls | 15 [5 to 19]

10. Other Pre Specified Outcome: Frequency of Missed Calls
Description: Online structured survey of number of missed calls since last survey
Time Frame: Assessed at 2, 4, 6, 8, 10, 12, 14, and 16 weeks; summed total missed phone calls at week 16 reported
Population: As pre-specified, we assessed and analyzed this variable in caregiver mentees only
Measure: Median (Inter-Quartile Range); unit: phone calls
Arm/Group | Caregiver Mentees
Number analyzed (Participants) | 28
phone calls | 1 [0 to 2.5]

11. Other Pre Specified Outcome: Dropout Rate of Mentors and Mentees, Respectively
Description: Proportion of mentors and mentees, respectively, not completing study per protocol
Time Frame: Sixteen weeks
Population: This outcome was not assessed in the focus group arm, as pre-specified.
Measure: Count of Participants; unit: Participants
Arm/Group | Peer Mentors | Caregiver Mentees
Number analyzed (Participants) | 30 | 30
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: Four months (sixteen weeks) of active peer mentoring
Arm/Group | Focus Group Participants | Peer Mentors | Caregiver Mentees
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/36 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/36 | 0/32
Other Adverse Events (participants affected / at risk) | 0/19 | 0/36 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT04649164/Prot_SAP_000.pdf